CLINICAL TRIAL: NCT01389375
Title: Instrumental Sealing of Arterial Puncture Site Closure Device Versus Manual Compression Trial
Acronym: ISAR-CLOSURE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GE IDE No. PCD00111
Record Dates: First submitted 2011-07-05; First posted 2011-07-08 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2014-07

CONDITIONS: Coronary Artery Disease
Keywords: Closure Device; Coronary Angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FemoSeal® (Experimental): Device: FemoSeal®
  Interventions: Device: FemoSeal®
- ExoSeal® (Experimental): Device: ExoSeal®
  Interventions: Device: ExoSeal®
- Manual compression (Active Comparator): Other: Manual compression
  Interventions: Other: Manual compression

INTERVENTIONS:
Device: FemoSeal® — Closure device for femoral artery access closure
  Arms: FemoSeal®
Device: ExoSeal® — Closure device for femoral artery access closure
  Arms: ExoSeal®
Other: Manual compression — Conventional manual compression
  Arms: Manual compression

SUMMARY:
Are novel vascular closure devices noninferior to manual compression regarding access site complications after coronary angiography?

DETAILED DESCRIPTION:
Vascular closure devices have been shown to be safe and effective in reducing the time to hemostasis and immobilization when compared to manual compression following coronary angiography. This effect is beneficial in patients presenting with chronic back pain, prostate enlargement, mental impairment or other disorders that preclude prolonged bed rest.

However, adequately powered large scale randomized trials with vascular closure devices remain a gap in the scientific literature.

This trial compares, in a randomised design two novel vascular closure devices (FemoSeal & ExoSeal) versus manual compression after coronary angiography. This study is aimed to investigate if novel vascular closure devices are noninferior to manual compression regarding access site complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient between 18 and 85 years of age
* Patients undergoing femoral access coronary angiography
* Access only with 6 F sheath
* Patient must be competent for providing informed written consent

Exclusion Criteria:

* Peripheral arterial occlusive disease
* Prior peripheral artery surgery
* Percutaneous coronary intervention
* Femoral access device closure in last 30 days
* Scheduled Coronary Angiography/Intervention within 90 days
* Critical limb ischemic
* Uncontrolled hypertension >220/110 mmHg
* Coagulopathy (bleeding disorder)
* Local infection
* Common femoral artery lumen diameter < 5 mm
* Allergy to absorbable suture
* Autoimmune Disease
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4524 (Actual)
Dates: Start 2011-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Composite of arterial access related complications | 30 days
  Composite of arterial access related complications, defined as the composite of:
  * Rate of ipsilateral groin hematomas with largest diameter exceeding 5 cm
  * Pseudoaneurysm
  * AV-Fistula
  * Major bleeding
  * Critical limb ischemia
  * Local infection
  * Surgical repair
  * Revascularisation

SECONDARY OUTCOMES:
Time to hemostasis, from sheath removal to complete hemostasis | 30 days
Device deployment failure | 30 days
Need for repeated manual compression after end of closure procedure | 30 days
Cost-benefit Analysis | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Linhardt, MD, Principal Investigator — Deutsches Herzzentrum München, Klinik für Herz- und Kreislauferkrankungen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Klinikum rechts der Isar, Munich

REFERENCES:
- [Background] Schulz-Schupke S, Helde S, Gewalt S, Ibrahim T, Linhardt M, Haas K, Hoppe K, Bottiger C, Groha P, Bradaric C, Schmidt R, Bott-Flugel L, Ott I, Goedel J, Byrne RA, Schneider S, Burgdorf C, Morath T, Kufner S, Joner M, Cassese S, Hoppmann P, Hengstenberg C, Pache J, Fusaro M, Massberg S, Mehilli J, Schunkert H, Laugwitz KL, Kastrati A; Instrumental Sealing of Arterial Puncture Site-CLOSURE Device vs Manual Compression (ISAR-CLOSURE) Trial Investigators. Comparison of vascular closure devices vs manual compression after femoral artery puncture: the ISAR-CLOSURE randomized clinical trial. JAMA. 2014 Nov 19;312(19):1981-7. doi: 10.1001/jama.2014.15305. PMID 25399273
- [Derived] Gewalt SM, Helde SM, Ibrahim T, Mayer K, Schmidt R, Bott-Flugel L, Hoppe K, Ott I, Hieber J, Morath T, Byrne RA, Kufner S, Cassese S, Hoppmann P, Fusaro M, Schunkert H, Laugwitz KL, Kastrati A, Schupke S; Instrumental Sealing of Arterial Puncture Site-CLOSURE Device Versus Manual Compression (ISAR-CLOSURE) Trial Investigators. Comparison of Vascular Closure Devices Versus Manual Compression After Femoral Artery Puncture in Women. Circ Cardiovasc Interv. 2018 Aug;11(8):e006074. doi: 10.1161/CIRCINTERVENTIONS.117.006074. PMID 30354782
- [Derived] Xhepa E, Byrne RA, Schulz S, Helde S, Gewalt S, Cassese S, Linhardt M, Ibrahim T, Mehilli J, Hoppe K, Grupp K, Kufner S, Bottiger C, Hoppmann P, Burgdorf C, Fusaro M, Ott I, Schneider S, Hengstenberg C, Schunkert H, Laugwitz KL, Kastrati A; ISAR-CLOSURE investigators. Rationale and design of a randomised clinical trial comparing vascular closure device and manual compression to achieve haemostasis after diagnostic coronary angiography: the Instrumental Sealing of ARterial puncture site - CLOSURE device versus manual compression (ISAR-CLOSURE) trial. EuroIntervention. 2014 Jun;10(2):198-203. doi: 10.4244/EIJV10I2A33. PMID 24952057